CLINICAL TRIAL: NCT03617809
Title: Prevention of Perioperative Hypothermia in Patients Submitted to Laparoscopic Urological Surgery
Brief Title: Perioperative Hypothermia in Patients Submitted to Laparoscopic Urological Surgery
Status: Completed | Type: Observational
Sponsor: Ángel Becerra (Other)
Collaborators: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Sponsor-Investigator, Ángel Becerra, MD, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: 2018-089-1
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Hypothermia; Anesthesia; Anesthesia; Adverse Effect; Peroperative Complication; Postoperative Complications; Surgical Site Infection; Temperature Change, Body
Keywords: Prewarming; Perioperative hypothermia; Esophageal thermometer
MeSH Terms: conditions — Hypothermia; Intraoperative Complications; Postoperative Complications; Surgical Wound Infection; Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prewarming: Active Prewarming will be performed using a forced-air blanket (WarmTouch lower body blanket, Covidien Ltd, Mansfield, USA) over the whole body and connected to a forced-air warmer (WarmTouch Model 5900, Covidien Ltd, Mansfield, USA). Patients will be warmed using a surgical blanket during the intraoperative period. Esophageal thermometer will be used to measure the temperature throughout the intraoperative period.
  Interventions: Procedure: Preoperative warming
- Control: Non-active prewarming. Patients will be warmed using a surgical blanket during the intraoperative period. Esophageal thermometer will be used to measure the temperature throughout the intraoperative period.

INTERVENTIONS:
Procedure: Preoperative warming — The prewarming time will not be decided by the clinical investigator. Prewarming time will depend on the time the patient has to wait before entering in the operating room.
  Groups: Prewarming

SUMMARY:
Hypothermia is a frequent perioperative complication. Its appearance can have deleterious effects such as perioperative bleeding or surgical site infection. Once the temperature has decreased, its treatment is difficult.

Preoperative warming prevents hypothermia, lowering the temperature gradient between core and peripheral compartments and reducing thermal redistribution. The most recent clinical practice guidelines advocate for active prewarming before induction of general anaesthesia since it is very effective in preventing perioperative hypothermia. However, the ideal warming time prior to the induction of anesthesia has long been investigated. This study aims to evaluate if different time periods of preoperative forced-air warming reduces the incidence of hypothermia at the end of surgery in patients submitted to laparoscopic urological surgery under general anesthesia. This is an observational prospective study comparing routine practice of pre-warming in consecutive surgical patients scheduled to laparoscopic prostatectomy or nephrectomy between August and December 2018. In this study 64 - 96 patients will be included and prewarming will be applied following routine clinical practice. The prewarming time will depend on the time the patient has to wait before entering in the operating theatre. Measurement of temperature will be performed using an esophagic thermometer. Patients will be followed throughout their hospital admission. Data will be recorded using a validated instrument and will be analysed using the statistics program R Core Team.

DETAILED DESCRIPTION:
Maintaining patient's temperature above 36 grades Celsius throughout the perioperative period is challenging. Thus, it is essential to monitor temperature in order to be able to take measures to avoid the appearance of hypothermia. Once the temperature has decreased, its treatment is difficult since the application of heat to the body surface takes a long time to reach the core thermal compartment. Intraoperative warming alone cannot avoid postoperative hypothermia. The application of forced-air warming system during the preoperative period has been shown to be the most effective measure to prevent hypothermia and maintain intraoperative normothermia. However, long time periods of prewarming would not be efficient. Thus, the ideal warming time prior to the induction of anesthesia has long been investigated.

Due to the searching of optimal prewarming time, the conductance of this study is justified.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic urological surgery under general anesthesia.

Exclusion Criteria:

* Active infection
* Intake of antipyretics within 24 hours before surgery
* Neuropathy
* Thyroid disorders
* Peripheral vascular disease
* Skin lesions
* History of hypersensitivity to skin contact devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective study comparing routine practice of prewarming in consecutive surgical patients scheduled to undergo elective laparoscopic urological surgery between August and December 2018. Ninety-nine patients will be included in this study and prewarming will be applied following routine clinical practice. The prewarming time will not be decided by the clinical investigator. Prewarming time will depend on the time the patient has to wait before entering in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Temperature | Through perioperative period, an average of 7 hours
  Asses the effect of prewarming in maintaining body temperature of patients undergoing elective laparoscopic urological surgery.
Temperature | From the arrival to the pre-anesthesia room to one hour after the arrival to the postanesthetic care unit an average of 7 hours.
  Differences in body core temperature throughout the perioperative period among different groups

SECONDARY OUTCOMES:
Surgical site infection | Through patient's stay in hospital, an average of 15 days
  Asses the effect of prewarming in preventing surgical site infection of patients undergoing elective laparoscopic urological surgery.
Postoperative shivering (using a dichotomous scale: yes or no) | Immediate postoperative period, an average of 1 hour.
  To assess the effect of prewarming in the prevalence of postoperative shivering of patients undergoing laparoscopic urological surgery.
Risk factors of perioperative hypothermia | Throughout the perioperative period, an average of 7 hours.
  To assess the effect of perioperative factors, related to the characteristics of patients and the surgery on provoking a greater drop of perioperative temperature.
Perioperative bleeding | Throughout the perioperative period, an average of 7 hours.
  Asses the effect of prewarming on decreasing perioperative bleeding of patients undergoing elective laparoscopic urological surgery.
Postoperative pain, using the visual analogue scale, from 0 to 10 | Immediate postoperative period, an average of 1 hour.
  Asses the effect of prewarming on decreasing postoperative pain of patients undergoing elective laparoscopic urological surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Becerra, MD, Principal Investigator — Doctor Negrin University Hospital
Locations (1):
- Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD are to be shared with other researchers when required once the study is completed and global data are published.